CLINICAL TRIAL: NCT07322484
Title: The Effect of Training Programs Based on Different Supportive Care Models in Childbirth on Midwifery Students' Clinical Self-Efficacy and Psychological Outcomes
Brief Title: Supportive Care-Based Training and Psychological Outcomes in Midwifery Students
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Gozde Gokce Isbir, Professor, Mersin University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AGY
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-09

CONDITIONS: Clinical Self-Efficacy; Psychological Outcomes; Secondary Traumatic Stress
Keywords: Trauma-Informed Care; Supportive Care Models in Childbirth; Midwifery Education; Clinical Self-Efficacy; Anxiety; Secondary traumatic stress
MeSH Terms: conditions — Compassion Fatigue; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Universal Continuous Supportive Care Model Training (Experimental): The first study group consisted of midwifery students enrolled in the Perinatal Health Practices I course during the fall semester. Following standard hospital orientation, students received Universal Continuous Supportive Care Model Training in childbirth, developed in line with the recommendations of Adams et al. The training lasted four hours, including one hour of theoretical instruction and three hours of practical application.
  The training focused on the core principles of universal continuous supportive care, their integration into clinical practice, and the use of a supportive care skills checklist. The 20-item checklist was developed by the researchers based on the literature to support students' self-evaluation of supportive care skills and included four domains: physical support, emotional support, education/information, and advocacy. Students were also encouraged to use a structured anamnesis form to plan individualized care.
  Interventions: Other: Universal Continuous Supportive Care Model Training
- Trauma-Informed Supportive Care Model Training (Experimental): The second study group consisted of midwifery students enrolled in the Perinatal Health Practices II course during the spring semester. Following standard hospital orientation, students received Trauma-Informed Supportive Care Model Training in childbirth, based on the recommendations of the Centre for Early Child Development. The training lasted four hours, including one hour of theoretical instruction and three hours of practical application.
  The training addressed the core principles of trauma-informed care, trauma-sensitive communication, and individualized care, with emphasis on integration into clinical practice. A 20-item trauma-informed supportive care checklist was introduced to support students' self-evaluation, structured around recognition and compassion, communication and collaboration, consistency and continuity, and understanding diversity. A trauma-informed anamnesis form was also used to guide individualized care planning.
  Interventions: Other: Trauma-Informed Supportive Care Model Training

INTERVENTIONS:
Other: Universal Continuous Supportive Care Model Training — The first study group consisted of midwifery students enrolled in the Perinatal Health Practices I course during the fall semester. Following standard hospital orientation, students received Universal Continuous Supportive Care Model Training in childbirth, developed in line with the recommendations of Adams et al. The training lasted four hours, including one hour of theoretical instruction and three hours of practical application.
  The training focused on the core principles of universal continuous supportive care, their integration into clinical practice, and the use of a supportive care skills checklist. The 20-item checklist was developed by the researchers based on the literature to support students' self-evaluation of supportive care skills and included four domains: physical support, emotional support, education/information, and advocacy. Students were also encouraged to use a structured anamnesis form to plan individualized care.
  Arms: Universal Continuous Supportive Care Model Training
Other: Trauma-Informed Supportive Care Model Training — The second study group consisted of midwifery students enrolled in the Perinatal Health Practices II course during the spring semester. Following standard hospital orientation, students received Trauma-Informed Supportive Care Model Training in childbirth, based on the recommendations of the Centre for Early Child Development. The training lasted four hours, including one hour of theoretical instruction and three hours of practical application.
  The training addressed the core principles of trauma-informed care, trauma-sensitive communication, and individualized care, with emphasis on integration into clinical practice. A 20-item trauma-informed supportive care checklist was introduced to support students' self-evaluation, structured around recognition and compassion, communication and collaboration, consistency and continuity, and understanding diversity. A trauma-informed anamnesis form was also used to guide individualized care planning.
  Arms: Trauma-Informed Supportive Care Model Training

SUMMARY:
The aim of this study is to comparatively evaluate the effects of trauma-informed supportive care model training in childbirth and universal supportive care model training in childbirth provided to midwifery students on their clinical skill self-efficacy in the delivery room, state anxiety, and secondary traumatic stress levels.

DETAILED DESCRIPTION:
This study was designed as a quasi-experimental comparative study. Data will be collected from fourth-year midwifery students enrolled in the Midwifery Department of Mersin University during the 2025-2026 academic year who undertake clinical practice in the delivery room of Mersin City Training and Research Hospital. Students who meet the inclusion criteria will be informed about the purpose and procedures of the study, and written informed consent will be obtained. Participants will be allocated to either the universal supportive care model training group or the trauma-informed supportive care model training group based on their academic semester (fall or spring), in line with the existing curriculum structure.

Both training programs will be delivered through theoretical and practical sessions prior to clinical application. Data will be collected from the participants themselves at three time points: before the intervention, immediately after providing childbirth care in the delivery room, and one week after the intervention, using validated self-report measurement tools assessing clinical skill self-efficacy, state and trait anxiety, and secondary traumatic stress levels. The planning, implementation, and reporting of the study will be conducted in accordance with relevant ethical principles and reporting guidelines for quasi-experimental research.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in the study
* Native Turkish speakers
* Enrollment as a fourth-year student in the Midwifery Department of Mersin University during the 2025-2026 academic year
* Enrollment in Perinatal Health Practices I or Perinatal Health Practices II
* Participation in delivery room clinical practice at Mersin City Training and Research Hospital
* No diagnosed psychiatric disorder and no use of psychiatric medication

Exclusion Criteria:

* Withdrawal from the study at any stage upon the participant's own request

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-07-08 (Estimated); Study Completion 2026-07-08 (Estimated)

PRIMARY OUTCOMES:
Clinical Skills Self-Efficacy | before the training and immediately after completion of delivery room clinical practice
  Midwifery students' clinical skills self-efficacy was assessed using the Clinical Skills Self-Efficacy Scale (CSSES). The scale was developed by Kang et al. (2019) to evaluate individuals' self-efficacy related to clinical practice. It consists of cognitive, affective, and psychomotor subdimensions. The Turkish version includes 11 items rated on a 5-point Likert scale ranging from 1 = strongly disagree to 5 = strongly agree, with higher scores indicating higher clinical self-efficacy. The Turkish adaptation demonstrated high internal consistency (Cronbach's alpha = .91).
State and Trait Anxiety | Trait Anxiety-before the training and one week after completion of delivery room practice; State Anxiety-immediately after completion of delivery room practice
  Midwifery students' anxiety levels were assessed using the State-Trait Anxiety Inventory (STAI), developed by Spielberger et al. (1970). The inventory consists of two subscales-State Anxiety and Trait Anxiety-each comprising 20 items rated on a 4-point Likert scale. Some positively worded items are reverse scored. Total scores reflect individuals' current (state) or general (trait) anxiety levels, with higher scores indicating higher anxiety. The Turkish version of the scale demonstrated high reliability, with Cronbach's alpha coefficients ranging from .94-.96 for the State Anxiety subscale and .83-.87 for the Trait Anxiety subscale.

SECONDARY OUTCOMES:
Secondary Traumatic Stress | Time Frame: one week after completion of delivery room clinical practice
  Midwifery students' secondary traumatic stress levels were assessed using the Secondary Traumatic Stress Scale (STSS), developed by Bride et al. (2005). The scale consists of 17 items across three subdimensions-avoidance, arousal, and intrusion-and is rated on a 5-point Likert scale. Total scores range from 17 to 85, with higher scores indicating higher levels of secondary traumatic stress. The Turkish version of the scale demonstrated high internal consistency, with a reported Cronbach's alpha coefficient of .91.

CONTACTS AND LOCATIONS:
Locations (1):
- Gozde Gokce Isbir, Mersin, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No